CLINICAL TRIAL: NCT03198819
Title: Powder Topical Rifampicin on Reducing Infections After Neural Tube Defect Surgery in Infants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, nihat demir, M.D, Yuzuncu Yil University
Record Dates: First submitted 2016-08-15; First posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Postoperative Infection Rates
Keywords: Topical rifampicin, neural tube defects, infection, newborn
MeSH Terms: conditions — Neural Tube Defects; Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Rifampisin group: Researchers will administer topical Rifampicin and intravenous cefotaxime
  1. For Rifampicin; 10 mg/kg/day, 24 h infusion on defect area during 3 days
  2. For cefotaxime; 50 mg/kg/day, twice a day, intravenous during 5 days.
  Interventions: Drug: Local Rifampisin and İnrtravenous cefotaxime
- Control group: Researchers will only administer intravenous cefotaxime
  1) Doses; 50 mg/kg/day, twice a day, intravenous during 5 days.
  Interventions: Drug: Local Rifampisin and İnrtravenous cefotaxime

INTERVENTIONS:
Drug: Local Rifampisin and İnrtravenous cefotaxime
  Other Names: Only intravenous cefotaxim

SUMMARY:
The correct timing and technique of neural tube defect (NTD) repairs significantly decreases the morbidity and mortality of NTD cases. However, infections related to the surgery are still common. We investigated the effects of topical rifampicin (RIF) combined with routine prophylaxis in newborns with open NTD.

DETAILED DESCRIPTION:
The study will be conducted in the Yuzuncu Yil University neonatal intensive care unit, Van, Turkey. The data of 60 neonates diagnosed with open NTD, who will be underwent surgical intervention between August 2016 and December 2017, will be prospectively evaluated. These cases will be randomised.These neonates are going to divide into two groups: the experimental group and the control group. The experimental group will be consisted of 30 newborns diagnosed with open NTDs, administered topical RIF (10 mg/kg/day, 24 h infusion) and cefotaxime (50 mg/kg/day, two doses, iv), and the control group will be consisted of 30 newborns diagnosed with open NTDs, administered cefotaxime (50 mg/kg/day, two doses).

In this study, researchers will be investigated whether prophylactic topical RIF applied on a pre-operative mesh in newborns with open NTD reduce the rate of SSIs and meningitis/ VP shunt infections after surgery. For deep incisional primary SSIs will be evaluated according to the diagnostic criteria of the United States (U.S.) Centers for Disease Control and Prevention (CDC) (1). The diagnosis of VP shunt infections will be made after extensive clinical and laboratory evaluations. the diagnosis of to make shunt infections, criteria of the Hydrocephalus Clinical Research Network (HCRN) will be taken into consideration (2).

Topical RIF Application Procedure The NTD site will be covered with a sterile gauze dressing in the first hours of life after birth in all babies with open NTDs. Then, 10 mg/kg/day RIF will be added to 24 ml of saline (0,9% NaCl), and this will be applied to the mesh as an infusion at a 1cc/h speed . Every day, the same dose of RIF will be delivered to the mesh,changed daily, as a 24-hour infusion until the patient could be operated. After the patient is operated, the RIF infusion delivered to the mesh will be stopped. The cefotaxime treatment will be continued until 72 hours post-op (3).

ELIGIBILITY:
Inclusion Criteria:

* Newborns who have open NTDs

Exclusion Criteria:

* Healthy newborns

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will be conducted in the Yuzuncu Yil University neonatal intensive care unit, Van, Turkey. The data of 60 neonates diagnosed with open NTD, who will be underwent surgical intervention between August 2016 and December 2017, will be prospectively evaluated. These cases will be randomised.These neonates are going to divide into two groups: the experimental group and the control group. The experimental group will be consisted of 30 newborns diagnosed with open NTDs, administered topical RIF (10 mg/kg/day, 24 h infusion) and cefotaxime (50 mg/kg/day, two doses, iv), and the control group will be consisted of 30 newborns diagnosed with open NTDs, administered cefotaxime (50 mg/kg/day, two doses).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Surgical site infections | within 30 days
  Deep incisional primary surgical site infections (SSIs) will be evaluated according to the diagnostic criteria of the United States (U.S.) Centers for Disease Control and Prevention (CDC). Accordingly, a diagnosis of infection will be established when fasciae, muscles or deep soft tissues associated with a surgical incision are affected within the first 30 postoperative days or when a foreign body (implant, etc.) leaves at the operation site will be observed within one year after the operation.
The diagnosis of ventriculoperitoneal (VP) shunt infection | within one month
  The diagnosis of VP shunt infections will be made after extensive clinical and laboratory evaluations. The diagnosis of to make shunt infections, criteria of the Hydrocephalus Clinical Research Network (HCRN) will be taken into consideration.
  Shunt infection will be defined as follows:
  1. the identification of organisms on a culture or Gram stain from cerebrospinal fluid (CSF), a wound swab or pseudocyst fluid;
  2. wound breakdown with visible shunt hardware;
  3. the presence of an abdominal pseudocyst (even in the absence of positive cultures); or
  4. positive blood cultures in a baby with a VP shunt.

SECONDARY OUTCOMES:
Length of hospitalization | within 6 months
  Researchers will evaluate as follows:
  1)Length of hospitalization,
  1)The cost of hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: nihat demir, Study Director — yüzüncüyıl üniversitesi
Locations (1):
- Yuzuncu yil medical school, Van, Outside of the US, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Garner JS, Jarvis WR, Emori TG, Horan TC, Hughes JM. CDC definitions for nosocomial infections, 1988. Am J Infect Control. 1988 Jun;16(3):128-40. doi: 10.1016/0196-6553(88)90053-3. PMID 2841893
- [Result] Beckman JM, Amankwah EK, Tetreault LL, Tuite GF. Reduction in CSF shunt infection over a 10-year period associated with the application of concentrated topical antibiotic powder directly to surgical wounds prior to closure. J Neurosurg Pediatr. 2015 Dec;16(6):648-61. doi: 10.3171/2014.12.PEDS13675. Epub 2015 Sep 18. PMID 26382185
- [Result] Demir N, Peker E, Gulsen I, Kocaman S, Tuncer O, Kirimi E. Powder Topical Rifampin for Reducing Infections After Neural Tube Defect Surgery in Infants. World Neurosurg. 2016 Nov;95:165-170. doi: 10.1016/j.wneu.2016.07.092. Epub 2016 Aug 6. PMID 27506408